CLINICAL TRIAL: NCT07014891
Title: A Study on Visual Feedback Motor Control Training Using Near-Infrared Spectroscopy (fNIRS) Brain Functional Imaging for Walking Function Recovery in Stroke Patients
Brief Title: fNIRS-Driven Visual Feedback Training to Restore Walking After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Xue Jiang, Associate Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024PS1843K
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: stroke; visual feedback; Functional near-infrared spectroscopy; walking ability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intelligent Visual Feedback Motor Control Training (Experimental): Patients receive motor control training using the Intelligent Visual Feedback Motor Control Training System (Monitored Rehab Systems B.V., 2031 CW Haarlem, The Netherlands), with the Monitored Rehab Systems-Functional Squat selected for training. The patient is in a supine position, with both feet fixed at the correct position on the pushing training board. The relative position of the patient is displayed on the computer screen. The system uses the height, length, and size of images to represent the degree of joint flexion/extension and the duration of muscle contraction, while the speed of moving images reflects the speed of joint movement and muscle contraction during exercise. Patients complete various simulated actions through interactive video games. The load of exercise training can be adjusted according to the patient's functional status and tolerance. The training is conducted once a day, 20 minutes each time, 5 times a week, for a total of 4 weeks.
  Interventions: Device: Intelligent Visual Feedback Motor Control Training
- Bobath Ball Training (Active Comparator): Bobath Ball Training Specific operations include: ① In the supine position, the heel controls the ball to move back and forth; ② In the supine position, both feet step on the ball to perform stepping movements, etc. The training is conducted 1 session daily, 20 minutes per session, 5 days per week, for a total of 4 weeks.
  Interventions: Device: Bobath Ball Training

INTERVENTIONS:
Device: Intelligent Visual Feedback Motor Control Training — Patients receive motor control training using the intelligent training system (Monitored Rehab Systems B.V., 2031 CW Haarlem, The Netherlands). The Monitored Rehab Systems-Functional Squat is selected for lower - limb motor control training. The patient assumes a supine position, with both feet fixed at the correct position on the pushing - training board. The relative position of the patient can be displayed on the computer screen. The system represents the degree of joint flexion and extension and the duration of muscle contraction through the height, length, and size of images, while the speed of moving images reflects the speed of joint movement during exercise. Patients complete various simulated actions through interactive video games. During the training, the load of exercise training can be adjusted according to the patient's functional status and tolerance. The training is conducted once a day, 20 minutes per session, five times a week, for a total of four weeks.
  Arms: Intelligent Visual Feedback Motor Control Training
Device: Bobath Ball Training — Bobath Ball Training Specific operations include: ① In the supine position, the heel controls the ball to move back and forth; ② In the supine position, both feet step on the ball to perform stepping movements, etc. The training is conducted 1 session daily, 20 minutes per session, 5 days per week, for a total of 4 weeks.
  Arms: Bobath Ball Training

SUMMARY:
The objective of this clinical trial is to investigate whether intelligent visual feedback-based lower limb motor control training is more effective than conventional rehabilitation training in promoting walking ability recovery among stroke patients with hemiplegia. The trial aims to address the primary question of the impact of intelligent visual feedback motor control training on the walking function of stroke patients with hemiplegia, and uses three-dimensional gait analysis for precise quantitative evaluation of therapeutic effects. Functional near-infrared spectroscopy (fNIRS) will be employed to explore patients' cerebral functional connectivity and cortical activation, and to analyze the correlation between fNIRS data and walking function scores (such as those from three-dimensional gait analysis), providing effective methods and a reliable reference basis for rehabilitation training of post-stroke hemiplegic patients.

Participants will be randomly divided into two groups: the experimental group receiving intelligent visual feedback motor control training, and the control group receiving Bobath ball training, 20 minutes per day, 5 days per week, for a total of four weeks. Before and after the treatment, indicators including fNIRS brain functional imaging, three-dimensional gait analysis, and Fugl-Meyer Assessment will be evaluated.

DETAILED DESCRIPTION:
Stroke is an injury with a high disability rate, and in recent years, it has shown a trend of younger onset. Its common complication is hemiplegia of one side of the body, which affects the walking stability and coordination of patients and severely impairs their quality of life. Exploring treatment measures that can improve the walking function of stroke patients is of great significance. Clinical studies have found that the decline in knee joint control ability in hemiplegic patients is a key problem leading to the decline in walking function. Traditional training mostly uses manual operations by therapists, with limited effects. Moreover, the single - rehabilitation treatment takes a long time and has a high training intensity, resulting in most patients developing negative emotions such as irritability and anger during the training process, and having poor compliance with rehabilitation training.

The MRS - FS (Monitored Rehab Systems-Functional Squat) system is a horizontal squat weight - reduction device that simulates the human squatting motion. Patients can safely perform early lower - limb strength training in a lying - down position. The real - time electronic images presented by this system help correct abnormal postures of patients, strengthen motor control, and thus improve walking function. In addition, the gamified and task - oriented exercise training mode can evoke positive emotions, improve patients' compliance with rehabilitation training, and enhance the effectiveness of exercise training. Existing studies have confirmed that MRS - FS can effectively improve lower - limb function, provide real - time feedback, improve knee joint control ability, and correct hemiplegic gait. However, currently, there are relatively few randomized controlled trial studies in clinical applications for the rehabilitation treatment of stroke patients with hemiplegia. Therefore, the treatment plan and efficacy evaluation of this system for stroke patients with hemiplegia are the key points for further exploration in this study.

Research shows that the main mechanism of functional recovery after stroke is the plastic change of the central nervous system and the remodeling of brain function. Functional near - infrared spectroscopy (fNIRS) is a non - invasive, safe, and non - invasive imaging technique. It can accurately measure the changes in cerebral cortex activity by detecting the changes in blood oxygen levels in the cerebral cortex. Different from technologies such as X - ray and CT, fNIRS does not involve ionizing radiation. This study innovatively uses fNIRS to explore the brain functional connectivity and activation status that are affected by intelligent visual feedback motor control training on patients' walking function, and further observes the recovery of brain function. At the same time, three - dimensional gait analysis is used to accurately quantify gait characteristics, providing an effective treatment method for the rehabilitation training of stroke patients with hemiplegia.

Research process: According to the inclusion and exclusion criteria, if a patient meets the enrollment conditions of this trial and agrees to participate in this study, after signing the informed consent form, they will start to enter this study. The study period is 4 weeks. Assessments will be conducted before treatment and 4 weeks after treatment, including: near - infrared brain function imaging; three - dimensional gait analysis; Fugl - Meyer Assessment - Lower Extremity. The treatment of patients may include intelligent visual feedback motor control training / Bobath ball training. Treatment grouping: Subjects will be randomly grouped, and each subject has an equal probability of being assigned to any group. There are two groups in total: Group A: Intelligent visual feedback motor control training (MRS - FS); Group B: Bobath ball training.

1. MRS - FS: The training includes six levels: random response, isometric contraction, random burst, control path, control position, and random deceleration. During the training process, the load of exercise training can be adjusted according to the patient's functional status and tolerance. It is carried out once a day, 20 minutes each time, 5 times a week, for a total of 4 weeks of treatment.
2. Bobath ball: Specifically, it includes: ①In the supine position, the heel controls the ball to move back and forth; ② In the supine position, both feet step on the ball to perform a stepping motion, etc. It is carried out once a day, 20 minutes each time, 5 times a week, for a total of 4 weeks of treatment. For the randomized study: Patients may be randomly assigned (like flipping a coin) to Group A or Group B. Assessments will be carried out before treatment and 4 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1: Vital signs are stable, with no severe cardiopulmonary diseases, making the patient suitable for exercise testing.

  2: All patients are diagnosed with stroke by head CT or MRI, with clinical manifestations of unilateral limb hemiplegia.

  3: The Brunnstrom stage of the lower limb is 3-5, quadriceps muscle strength is ≥ grade 3, modified Ashworth scale for the lower limb is < grade 2, and Hoffer walking scale is ≥ grade 2.

  4: This is their first onset of the disease, with a disease course of ≤ 6 months, and the condition is stable.

  5: Patients have no severe cognitive impairment or sensory aphasia, can understand and actively participate in the training program, and have provided informed consent by signing the consent form for this clinical study.

  6: Age: 18-75 years old, no gender restrictions.

Exclusion Criteria:

* 1: Patients with tumors, tuberculosis, hematological diseases, or functional impairments of vital organs such as the heart or liver.

  2: Those with lower limb musculoskeletal disorders, such as knee arthritis or lower limb fractures.

  3: Individuals with severe abnormal muscle tone in the limbs or joint contracture deformities.

  4: Patients experiencing severe pain that prevents them from tolerating physical activity.

  5: Special populations, such as individuals with mental illnesses, breastfeeding women, or pregnant women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy | Baseline, 4-weeks treatment
  Near-infrared Brain Functional Imaging：The testing areas cover the bilateral prefrontal lobes, motor areas, occipital lobes, and other brain regions. Within 1 week before treatment initiation, a physician will collect resting-state and task-state fNIRS data from enrolled patients.Resting-State Data Collection：The patient is fitted with an fNIRS measurement headcap. In a quiet, comfortable environment, they are instructed to sit, relax, keep eyes closed (without falling asleep), and data are collected for 5 minutes.Task-State Data Collection：A walking paradigm is set up. The test includes a 10-second preparatory phase where the patient stands at rest, followed by the task phase:Upon the command "Please start walking," the subject alternates stepping for 30 seconds.At the command "Stop," they cease walking and stand in place to rest for 30 seconds.
  This "walk-rest" cycle is repeated 4 times.Identical data collection will be completed within 1 week after treatment concludes.
Three-Dimensional Gait | Baseline, 4-weeks treatment
  * Gait spatiotemporal parameters
  * Lower limb joint angles
  * Lower limb joint moments
  * Ground reaction forces etc.

SECONDARY OUTCOMES:
Fugl Meyer Assessment | Baseline, 4-weeks treatment
  The Fugl-Meyer Assessment (FMA) is used to evaluate the lower limb motor function and coordination of research subjects. Modified from the Brunnstrom evaluation method, this scale is divided into two parts: upper limb and lower limb motor function assessment, with only the lower limb subscale (FMA-LE) applied in this study. The FMA-LE consists of 17 items, each graded into three levels (0 points = unable to perform; 1 point = partially performed; 2 points = fully performed), with a total score ranging from 0 to 34. A higher score indicates better lower limb motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Jiang, Study Chair — Shengjing Hospital
Locations (1):
- Rehabilitation Center of Shengjing Hospital, China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available under reasonable request after publication. Data will include de-identified participant data and the data dictionary. Requests can be submitted to the corresponding author. Request will be analyzed and ethical and legal implications of data sharing will be considered. Data will be shared after consent of study participants
Time Frame: After publication under reasonable request.

REFERENCES:
- [Result] Ferrari M, Quaresima V. A brief review on the history of human functional near-infrared spectroscopy (fNIRS) development and fields of application. Neuroimage. 2012 Nov 1;63(2):921-35. doi: 10.1016/j.neuroimage.2012.03.049. Epub 2012 Mar 28. PMID 22510258
- [Result] Lin CH, Chou LW, Luo HJ, Tsai PY, Lieu FK, Chiang SL, Sung WH. Effects of Computer-Aided Interlimb Force Coupling Training on Paretic Hand and Arm Motor Control following Chronic Stroke: A Randomized Controlled Trial. PLoS One. 2015 Jul 20;10(7):e0131048. doi: 10.1371/journal.pone.0131048. eCollection 2015. PMID 26193492
- [Result] Takahashi MTC, Balardin JB, Bazan PR, Boasquevisque DS, Amaro Junior E, Conforto AB. Effect of transcranial direct current stimulation in the initial weeks post-stroke: a pilot randomized study. Einstein (Sao Paulo). 2024 Jun 24;22:eAO0450. doi: 10.31744/einstein_journal/2024AO0450. eCollection 2024. PMID 38922218
- [Result] Cohen EJ, Quarta E, Bravi R, Granato A, Minciacchi D. Neural plasticity and network remodeling: From concepts to pathology. Neuroscience. 2017 Mar 6;344:326-345. doi: 10.1016/j.neuroscience.2016.12.048. Epub 2017 Jan 7. PMID 28069532
- [Result] Schnautz LS. Critical Care Nursing Clinics of North America. Cardiovascular disease in women. Preface. Crit Care Nurs Clin North Am. 2008 Sep;20(3):xi-xii. doi: 10.1016/j.ccell.2008.03.015. No abstract available. PMID 18644505
- [Result] Jarvis HL, Brown SJ, Price M, Butterworth C, Groenevelt R, Jackson K, Walker L, Rees N, Clayton A, Reeves ND. Return to Employment After Stroke in Young Adults: How Important Is the Speed and Energy Cost of Walking? Stroke. 2019 Nov;50(11):3198-3204. doi: 10.1161/STROKEAHA.119.025614. Epub 2019 Sep 26. PMID 31554503